CLINICAL TRIAL: NCT03510260
Title: Electronic Confirmed Versus Conventional Consenting Process (ECCCO)
Brief Title: Electronic Confirmed Versus Conventional Consenting Process: A Randomized Controlled Trial
Acronym: ECCCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-0063
Record Dates: First submitted 2018-04-16; First posted 2018-04-27 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Satisfaction; Risk Reduction
Keywords: Cesarean, Consent, Electronic, Satisfaction
MeSH Terms: conditions — Personal Satisfaction; Risk Reduction Behavior | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Unblinded randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Placebo Comparator): Subject will undergo regular consenting only. At our unit consent for an elective cesarean delivery occurs in the same day of surgery, few hours before the procedure in a private room in labor and delivery while awaiting surgery. The COMRADE questionnaire (our primary outcome) will be obtained after the completion of the paper consent form.
  Interventions: Other: Control Group
- Study Group I (Experimental): Subject will receive an electronic invitation to complete the consent process electronically and will proceed through the Confirmed Consent system prior to arrival to labor and delivery on day of surgery, which is the routine patient flow at this time. The COMRADE questionnaire (our primary outcome) will be obtained prior to the initiation of the traditional consent (as in control group) before the completion of the paper consent form, in order to assess satisfaction and understanding of the e-confirmed consenting process completed before the procedure. After completion of the survey, the subject will sign the regular paper consent for the procedure as standard in our institution.
  Interventions: Other: Study Group I
- Study Group II (Experimental): Subject will undergo the same intervention as group II but the COMRADE survey questionnaire will be obtained after the paper consent is obtained in order to assess whether both methods combined together improve the subjects' satisfaction of the consenting methods and better understanding of the surgical procedure.
  Interventions: Other: Study Group II

INTERVENTIONS:
Other: Study Group I — Study group I (e-confirmed consent only) will receive an electronic invitation to complete the consent process electronically.The COMRADE questionnaire (our primary outcome) will be obtained prior to the initiation of the traditional consent (as in control group).
  Other Names: e-confirmed consent
  Arms: Study Group I
Other: Study Group II — The study group II will undergo the same intervention as group II but the COMRADE survey questionnaire will be obtained after the paper consent
  Other Names: e-confirmed consent plus paper consent
  Arms: Study Group II
Other: Control Group — Subject will go through the consenting process at the day of surgery at the preop visit as standard in our institution only.
  Other Names: Standard paper consent only
  Arms: Control Group

SUMMARY:
· The target population for our study is women who present in their last clinic visit before delivery and are scheduled for an elective cesarean section. In that visit, the provider will notify the research team in order for the subject to be screened for the study. If the subject consents to participation, written informed consent will be obtained by person-to-person contact. The PI, study coordinator, or a collaborator will be responsible for the informed consent. After in-formed consent is obtained, the patient will be randomized to the following study groups:

The control group will undergo regular consenting only.

Study group I (e-confirmed consent only) will receive an electronic invitation to complete the consent process electronically and will proceed through the Confirmed Consent system prior to arrival to labor and delivery on day of surgery, which is the routine patient flow at this time. After completion of the survey, the subject will sign the regular paper consent for the procedure as standard in our institution.

The study group II will undergo the same intervention as group II but the COMRADE survey questionnaire will be obtained by phone or in person after the completion of the paper consent form.

DETAILED DESCRIPTION:
4.1 Screening, Recruitment, and Consenting:

* Under the direction of the PI, trained research staff will be available 24/7 to screen and con-sent patients according to study protocol. Patients will be enrolled at the time a decision for planned repeat cesarean after VBAC counseling is made in clinic.
* After informed consent is obtained, the patient will be randomized to the study group or the control group. A screening log will be used to track all patients approached for the study. Women will only be randomized in clinic.
* Recruitment: We will recruit all pregnant patient's decision was made for scheduled cesarean after VBAC counseling made by their managing clinical team who do not meet any of the ex-clusion criteria listed below. Once the inclusion criteria for our study are met, the primary team will inform the patient about the study and ask her authorization to contact one of the study personnel.
* Consenting process: Written consent will be obtained by direct person-to-person contact. The principal investigator, study coordinator, or a collaborator will be responsible for the informed consent. Non-English-speaking subjects are anticipated to be part of the study population and informed consent will be provided in their primary language.

The data collected will not be used for clinical diagnosis or treatment purposes.

Subjects will be reassured that participation in the study is voluntary and will not interfere with diag-nose or treatment of her condition.

The subjects will receive the same care and expertise as any other patient treated in our institution.

4.2. Randomization and Masking A confidential computer-generated simple randomization scheme (using STATA 14, Dallas, TX) will be prepared and provided on an ongoing basis to our study coordinator. A randomization log with group assignment, subject name, and medical record number will be used to track the randomization process.

The subject will be included in the analysis by intent-to-treat once the randomization assignment has been made.

4.3. Interventions The control group will undergo regular consenting only. At our unit consent for an elective ce-sarean delivery occurs in the same day of surgery, few hours before the procedure in a private room in labor and delivery while awaiting surgery. The COMRADE questionnaire (our primary outcome) will be obtained after the completion of the paper consent form.

Study group I (e-confirmed consent only) will receive an electronic invitation to complete the consent process electronically and will proceed through the Confirmed Consent system prior to arrival to labor and delivery on day of surgery, which is the routine patient flow at this time. The COMRADE questionnaire (our primary outcome) will be obtained prior to the initiation of the traditional consent (as in control group) before the completion of the paper consent form, in order to assess satisfaction and understanding of the e-confirmed consenting process completed before the procedure. After completion of the survey, the subject will sign the regular paper consent for the procedure as standard in our institution.

The study group II will undergo the same intervention as group II but the COMRADE survey questionnaire will be obtained after the paper consent is obtained in order to assess whether both methods combined together improve the subjects' satisfaction of the consenting methods and better understanding of the surgical procedure.

4.4. Survey Collection This is our primary outcome. Before the subject has the procedure, our research staff will be collecting a survey assessing understanding of procedure and satisfaction, please see attached survey with appli-cation. This survey will be obtained according to the interventions detailed in sections 3 & 4.3

ELIGIBILITY:
Inclusion Criteria:

* Women >18 and <50
* Plan for scheduled elective Cesarean
* English speaking

Exclusion Criteria:

* Patient unwilling or unable to provide consent
* Incarcerated patients
* Unable to complete e-confirmed consent (not able to access the confirmed consent from home)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Obstetrical population
Enrollment: 105 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
COMRADE Questionnaire | Up to 7 days after delivery
  a survey assessing understanding of procedure and satisfaction,

SECONDARY OUTCOMES:
Understanding Survey | Up to 7 days after delivery
  Survey or questionnaire to assess subject's understanding of the planned procedure

CONTACTS AND LOCATIONS:
Locations (1):
- UTMB Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No